CLINICAL TRIAL: NCT06636019
Title: Change in Choroidal Thickness of Myopic Eyes With a Myopia Control Contact Lens
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Augsburg (Other)
Responsible Party: Principal Investigator, Dr. med.Isabella Baur, Principal Investigator, University Hospital Augsburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-0398
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Myopia
Keywords: Myopia; Contact Lens; Myopia progression
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional arm (Experimental): The myopia control contact lens will be administered in this group.
  Interventions: Device: Myopia control contact lens

INTERVENTIONS:
Device: Myopia control contact lens — Myopia control contact lens is placed on the study eye.

SUMMARY:
In this study, the direct effect of the MiSight contact lens (Cooper Vision), a daily disposable contact lens recently approved in Germany for the treatment of myopia, will be investigated. The aim of this study is to demonstrate an increase in choroidal thickness due to the myopic defocus induced by the contact lens. The increase in choroidal thickness after 30 minutes of exposure to the myopic defocus induced by the contact lens will be demonstrated by measuring the subfoveal and macular choroidal thickness.

DETAILED DESCRIPTION:
The increasing incidence of short-sightedness (myopia) worldwide has led to the development of various therapies to control axial length myopia. The latest developments include contact lenses to inhibit the growth of the bulb length, which should influence the growth of the eye in childhood and adolescence by inducing a myopic defocus in the periphery of the retina.

In this study, the direct effect of the MiSight contact lens (Cooper Vision), a daily disposable contact lens recently approved in Germany for the treatment of myopia, will be investigated. The aim of this study is to demonstrate an increase in choroidal thickness due to the myopic defocus induced by the contact lens. The increase in choroidal thickness after 30 minutes of exposure to the myopic defocus induced by the contact lens will be demonstrated by measuring the subfoveal and macular choroidal thickness. In addition, the influence of accommodation will be investigated by measuring the choroidal thickness after 30 minutes of activity at near and far distance. One eye of each of 8 healthy subjects with myopic refraction from -0.5 diopters in the spherical equivalent will be included, with laterality (right/left) being randomized. The choroidal thickness is measured using optical coherence tomography (OCT), which is standard in clinical routine. The examination is non-invasive and is carried out at three points in time: The baseline measurement is carried out before inserting the contact lens, then after 30 minutes of exposure and near focusing. A further measurement is carried out within a week after a further 30 minutes of exposure and distance focusing, so that the results are not distorted by the previous near work. In addition, the axial length is determined at each of the 3 measurement times using optical biometry.

ELIGIBILITY:
Inclusion Criteria:

* myopic refraction
* consent to participate
* minimum age 18 years
* full legal capacity

Exclusion Criteria:

* ocular disease affecting imaging quality including but not limited to cataract, keratoconus
* ocular disease affecting choroidal thickness (pachychoroidal disease)
* astigmatism greater than 1,5 diopters
* best corrected distance visual acuity of 0,1 logMAR or worse
* status post eye surgery
* status post treatment for myopia control

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Choroidal thickness | 30 minutes
  Choroidal thickness is measured after contact lens wear.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Augsburg, Augsburg, Germany

IPD SHARING:
Plan to Share IPD: No